CLINICAL TRIAL: NCT06094257
Title: Prospective Cohort Study Comparing Sensory Outcome, Development of Chronic Pain and Phantom Pain, as Well as Patient Satisfaction in Cancer and Transgender Patients Undergoing Mastectomy and Reconstruction With and Without Reinnervation.
Brief Title: Prospective Study of Sensation and Satisfaction in Cancer and Transgender Mastectomy Patients
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22-09025293
Record Dates: First submitted 2023-10-03; First posted 2023-10-23 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Sensation Disorders; Sensation, Phantom; Pain, Postoperative; Pain, Chronic; Numbness; Sensory Disorder; Sensory Defect; Phantom Pain; Phantom Sensation
Keywords: Sensation; Reinnervation; Peripheral nerve; Reconstruction; Breast reinnervation; Chest reinnervation; Gender-affirming mastectomy; Breast reconstruction; Peripheral nerve repair; Targeted nipple areolar complex; Targeted nipple areolar complex reinnervation
MeSH Terms: conditions — Sensation Disorders; Phantom Limb; Pain, Postoperative; Chronic Pain; Hypesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Nipple sparing mastectomy (NSM) and implant reconstruction: Nipple sparing mastectomy (NSM) and implant reconstruction
  Interventions: Diagnostic Test: Sensory testing
- Nipple sparing mastectomy (NSM) and autologous reconstruction: Nipple sparing mastectomy (NSM) and autologous reconstruction
  Interventions: Diagnostic Test: Sensory testing
- Gender mastectomy with free nipple grafting: Gender mastectomy with free nipple grafting
  Interventions: Diagnostic Test: Sensory testing
- Control patients matched by surgical procedure, age, BMI and mastectomy weight.: Control patients matched by surgical procedure, age, BMI and mastectomy weight.
  Interventions: Diagnostic Test: Sensory testing

INTERVENTIONS:
Diagnostic Test: Sensory testing — Quantitative sensory testing (QST) will be performed. QST was developed to standardize the noninvasive assessment of the somatosensory nervous system and quantify functioning of all aspects of sensation (light touch, pressure, warm, cold, pain, vibration): 1. Thermal detection (Medoc TSA system): Cold detection threshold B) Warm detection threshold C) Heat pain threshold 2. Mechanical detection threshold (MRC Opti Hair von Frey Filaments) 3. Two-point discrimination (MRC Opti Hair von Frey Filaments) 4. Mechanical pain threshold (MRC Pinprick Stimulator) 5. Pressure pain threshold (Medoc Pressure algometer) 6. Tinel sign on physical exam 7. Vibration (tuning fork)

SUMMARY:
During breast surgery, sensory nerves are cut which may lead to reduced sensation and pain. Surgical reinnervation techniques have been developed with the aim of improving postoperative sensation by preserving the nerves and connecting them to the nipple and areola. The investigators aim to compare postoperative sensation and patient reported outcomes in patients undergoing reinnervation versus those not undergoing reinnervation to determine if there is a difference. The investigators will investigate this in patients undergoing gender-affirming mastectomy, implant-based breast reconstruction and autologous breast reconstruction. The investigators will use various tools that measure sensation quantitatively.

DETAILED DESCRIPTION:
SIGNIFICANCE

During removal of breast tissue that is required for mastectomy procedures, the nerves that supply the breast skin and the nipple areola complex (NAC) are sacrificed. This results in fair to poor sensation in 50-90% of patients, decreased patient satisfaction and increased risk of injury. Further, when nerves are transected, axons sprout from the proximal free nerve end and form neuromas that cause chronic pain (CP) and phantom pain (PP) in ~60% and 30-80% of patients, respectively. With the implementation of advanced peripheral nerve surgery techniques, it has become possible to preserve, transfer and graft nerves to the insensate areas of the reconstructed breast/chest to provide sensation in cancer and transgender patients. Multiple studies have shown increased patient satisfaction and sensation after reinnervation as compared to no reinnervation. However, there are several limitations to currently published clinical outcome studies: 1)Lack of comprehensive objective outcome measures to test all aspects of the somatosensory nervous system. No study to date has utilized the protocol for Quantitative Sensory Testing (QST) that was developed by the German Research Network on Neuropathic Pain (DFNS) and provides a validated and standardized approach to test all nociceptive and non- nociceptive sensory functions including small unmyelinated C fibers, myelinated A-alpha, A-beta, and A-delta fibers. This comprehensive, standardized and validated approach has been adopted internationally to evaluate sensory conditions and allows for objective outcome assessment and comparison. 2)Gap in knowledge regarding reinnervation outcomes after implant- based reconstruction. Most sensory studies were performed in patients undergoing autologous reconstruction with only few studies discussing reinnervation in the context of implant- based breast reconstruction. However, the most common type of reconstruction after breast cancer remains implant based reconstruction accounting for 80% of breast reconstruction cases. Therefore, it is important to investigate this population further to determine whether reinnervation is successful and should be offered to this patient population. 3)Limited understanding of sensory outcome after transgender mastectomy. Sensory outcome is important to >90% of patients undergoing transgender mastectomy with free nipple grafting (FNG), which is the most common procedure performed in transgender patients. Our team has described chest reinnervation in this patient population with good sensory outcomes. However, a prospective clinical trial with comprehensive outcome measurements including QST and patient reported outcome measures (PROMs) with control group is required to further examine the role of reinnervation in transgender chest surgery. 4)Insufficient prospective data on PP and CP. There are very few prospective studies reporting the incidence of PP and CP after cancer and transgender mastectomy and the results are inconsistent. Further, the percentage of chronic breast/chest pain patients with true neuropathic pain (NP) is unclear. In addition, although we know from other patient populations (amputees) that nerve reconstruction significantly decreases the incidence of CP and PP, there is no data on whether breast reinnervation influences the percentage of patients who will develop these conditions. 5)Prospective comparison of reinnervation outcomes between autologous reconstruction, implant reconstruction and gender mastectomy has not been performed. Breast reinnervation has rapidly evolved and is becoming a widely employed addition to breast and chest reconstruction. However, it remains unclear how these patient populations compare, and which patients obtain good sensory outcome warranting the longer operative times and higher cost of reinnervation.

The broad objective of this proposal is to prospectively compare objective data on sensory outcomes using QST and PROMs in patients undergoing reinnervation after A) nipple sparing mastectomy (NSM) and implant reconstruction B) NSM and autologous reconstruction C) gender mastectomy with FNG and D) control patients matched by surgical procedure, age, BMI and mastectomy weight. This preliminary data will be used to apply for government funding (NIH K23) to conduct a randomized controlled multi- center clinical trial to evaluate reinnervation versus no reinnervation after mastectomy in cancer and transgender care. The objectives of this larger scale study are to A) obtain objective QST sensory measurements and PROM outcomes across institutions, B) determine the chances of reinnervation success based on variables such as patient factors (age, comorbidities, adjuvant treatment), mastectomy factors (incision type, mastectomy weight), breast reconstruction techniques (retropectoral, prepectoral, direct- to implant, expander reconstruction, implant size, implant type, types of autologous reconstruction), chest reconstruction techniques and nerve transfer techniques (number of nerves, length of allograft, size of allograft etc.) C) perform a cost- benefit analysis and D) develop evidence-based guidelines for breast/ chest reinnervation after mastectomy.

SPECIFIC AIMS

All aims will analyze and compare the following patient groups: a) NSM and implant reconstruction with reinnervation b) NSM with autologous reconstruction with reinnervation c) gender mastectomy with FNG with reinnervation d) controls matched by surgical procedure (implant, autologous, transgender), BMI, age, gender and mastectomy weight.

Aim 1A: Analysis of all aspects of sensation with QST. Aim 1B: Evaluation of timing of return of sensation. Aim 2: Assessment of CP and PP. Aim 3: Analysis of patient satisfaction.

HYPOTHESIS

Breast reinnervation does not improve sensation/patient satisfaction as compared to mastectomy with no reinnervation. Further, there is no difference in prevalence of CP and PP.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patient is scheduled for gender mastectomy surgery (including nipple sparing mastectomy and mastectomy with free nipple graft) or NSM with breast implant or autologous reconstruction
* Patient is capable and willing to provide informed consent

Exclusion Criteria:

* Patient has a nerve condition that does not allow for assessment of sensation
* Any subject who at the discretion of the Investigator is not suitable for inclusion in the study or is unlikely to comply with follow-up schedule
* Currently prescribed medication known to impact nerve regeneration or to cause peripheral neuropathy
* Bilateral reconstruction with non-uniform treatment (i.e. 1 reconstructed breast is non-neurotized, 1 reconstructed breast is neurotized)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Massachusetts General Hospital (MGH) and Weill Cornell Medicine (WCM) are ideally suited for enrollment of patients in this study. Both institutions are high-volume center of expertise for gender affirming mastectomy and breast reconstructions as well as peripheral nerve surgery.
  Patients will be matched by BMI, age and mastectomy weight. Patients scheduled to undergo gender affirming mastectomy or breast reduction surgery at MGH and WCM will be evaluated for the study and will be presented with the option to hear about the study by our research assistant. Those interested in the study will be presented with all the necessary details required by the IRB including a study fact sheet. Verbal consent will be obtained and documented.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Change in Breast Q scores | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  All BREAST-Q scores range from 0-100. The scores are computed from the responses to the separate questions by adding them together and converting the score to a scale from 0 to 100 (similar to conversion into a percentage). A higher score means high satisfaction or better health-related quality of life.
Change in Gender-Q scores | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  All Gender-Q scores range from 0-100. The scores are computed from the responses to the separate questions by adding them together and converting the score to a scale from 0 to 100 (similar to conversion into a percentage). A higher score means high satisfaction or better health-related quality of life.
Change in cold detection threshold | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Thermal detection measured by Medoc TSA system
Change in warm detection threshold | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Thermal detection measured by Medoc TSA system
Change in heat pain threshold | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Thermal detection measured by Medoc TSA system
Change in mechanical detection threshold | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Measured by MRC Opti Hair von Frey Filaments
Change in two-point discrimination | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Measured by MRC Opti Hair von Frey Filaments
Change in mechanical pain threshold | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Measured by MRC Pinprick Stimulator
Change in pressure pain threshold | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Measured by Medoc Pressure algometer
Change in Tinel sensation | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Measure on physical exam
Change in vibration sensation | preoperative, postoperative at 1 month, 3 months, 6 months, and 1 year
  Measured by tuning fork

SECONDARY OUTCOMES:
Change in Breast Q scores long term | Annually at 2-10 years post-operation
  All BREAST-Q scores range from 0-100. The scores are computed from the responses to the separate questions by adding them together and converting the score to a scale from 0 to 100 (similar to conversion into a percentage). A higher score means high satisfaction or better health-related quality of life.
Change in Gender Q scores long term | Annually at 2-10 years post-operation
  All Gender-Q scores range from 0-100. The scores are computed from the responses to the separate questions by adding them together and converting the score to a scale from 0 to 100 (similar to conversion into a percentage). A higher score means high satisfaction or better health-related quality of life.
Change in vibration sensation | Annually at 2-10 years post-operation
  Measured by tuning fork
Change in Tinel sensation | Annually at 2-10 years post-operation
  Measure on physical exam
Change in pressure pain threshold | Annually at 2-10 years post-operation
  Measured by Medoc Pressure algometer
Change in mechanical pain threshold | Annually at 2-10 years post-operation
  Measured by MRC Pinprick Stimulator
Change in two-point discrimination | Annually at 2-10 years post-operation
  Measured by MRC Opti Hair von Frey Filaments
Change in mechanical detection threshold | Annually at 2-10 years post-operation
  Measured by MRC Opti Hair von Frey Filaments
Change in heat pain threshold | Annually at 2-10 years post-operation
  Thermal detection measured by Medoc TSA system
Change in warm detection threshold | Annually at 2-10 years post-operation
  Thermal detection measured by Medoc TSA system
Change in cold detection threshold | Annually at 2-10 years post-operation
  Thermal detection measured by Medoc TSA system

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Gfrerer, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided